CLINICAL TRIAL: NCT03785431
Title: Vascular Healing Pattern, Vasoreactivity, and Quality of Life in Patients With ST Segment Elevation Myocardial Infarction Treated With Primary Percutaneous Coronary Intervention With Sirolimus Eluting FANTOM Bioresorbable Vascular Scaffold With Long Term Clinical, Near Infrared Spectroscopy and Optical Coherence Tomography Follow-up: A FANTOM STEMI Pilot Study
Brief Title: Vascular Healing After Implantation of FANTOM Bioresorbable Scaffold in STEMI: A FANTOM STEMI Study
Acronym: FANTOM STEMI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Łukasz Kołtowski, Adjunct Prof., MD, PhD, Medical University of Warsaw
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KB/169/2016
Record Dates: First submitted 2018-11-13; First posted 2018-12-24 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: STEMI; Cardiovascular Disease; Bioresorbable Scaffold
Keywords: STEMI; cardiovascular disease; bioresorbable scaffold
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Cardiovascular Diseases | interventions — Percutaneous Coronary Intervention; Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Patient diagnosed with ST elevation myocardial infarction will undergo bioresorbable stent deployment in culprit lesion.
  Interventions: Device: PCI with Phantom Bioresorbable Scaffold

INTERVENTIONS:
Device: PCI with Phantom Bioresorbable Scaffold — Once baseline angiography is performed and all eligibility criteria are met, the patient is included in the study. The target lesion should be crossed with a standard coronary guidewire. Next, the NIRS/IVUS and OCT probe is inserted and a pullback is being performed to evaluate the lesion and vessel morphology. The predilatation with 1:1 non-compliant or semi-compliant balloon is mandatory. Thereafter the scaffold should be inserted and position across the target lesion. Lesions up to 14 mm should be covered with the 18 mm device, for lesions of 15-20 mm a 24 mm device should be used. The scaffold will be deployed with intent to achieve the inner diameter to the reference vessel ration of 1:1 using a single inflation. Post-dilatation using a non-compliant balloon should be performed to achieve complete scaffold apposition and reduce the residual angiographic stenosis below 20%. The final NIRS/IVUS and OCT of the target vessel should be performed.
  Other Names: OCT and NIRS-IVUS Evaluation

SUMMARY:
The study will assess the safety and performance of the Fantom sirolimus eluting bioresorbable vascular scaffold (BVS) in the acute setting of myocardial infarction with unstable lesions and thrombogenic milieu.This is a prospective evaluation of clinical and patient related measures in STEMI patient who undergo urgent primary percutaneous coronary intervention (PCI) with stent implantation. Patients with culprit lesions with 2.5 - 3.5 mm diameter and located in one of the main coronary arteries will be included in the trial and prospectively observed. The study will comprise 20 patients, who will undergo additional evaluation with optical coherence tomography (OCT) and near-infrared spectroscopy/intravascular ultrasound (NIRS/IVUS) at baseline, 6 months, 18-24 months and 36 months. The device will be delivered in sizes 2.5 and 3.0 in diameter / 18 and 24 mm and 3.5 mm x 18 mm in length.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the acute safety and feasibility of implantation of the sirolimus-eluting bioresorbable Fantom scaffold BVS in the setting of ST segment elevation myocardial infarction (STEMI), as well as the mid and long-term clinical efficacy and healing pattern of the device, the plaque modification and patient related outcomes, including quality of life and patient preferences.

Primary end-point

* Procedural success defined as acute angiographic success (residual stenosis <20% and Thrombolysis In Myocardial Infarction (TIMI) flow 3) without in-hospital major adverse cardiac events (MACE) (19) Secondary end-points
* Angiographic success defined as device implantation into target lesion with residual stenosis of < 20% and presence of grade 3 TIMI flow assessed by angiography. (19)
* Quantitative coronary angiographic measurements including minimum lumen diameter (mm), diameter stenosis (%), late lumen loss (mm), evaluated post-procedure, at 6, 18 and 36 months
* OCT measurements at patient level including mean lumen area (mm2), mean scaffold area (mm2), mean vessel area (mm2), mean/min./max. neointima thickness (μm), neointima area (mm2), scaffold area obstruction (%), symmetry of the neointima thickness, malposed strut ratio (%), malposed strut total (n), mean malposition distance (mm), malposition area (mm2) evaluated post-procedure, at 6, 18 and 36 months (16)
* OCT measurements at scaffold level including mean lumen area (mm2), mean scaffold area (mm2), mean vessel area (mm2), mean/min./max. neointima thickness (μm), neointima area (mm2), scaffold area obstruction (%), symmetry of the neointima thickness, malposed strut ratio (%), malposed strut total (n), mean malposition distance (mm), malposition area (mm2) evaluated post-procedure, at 12, 24 and 36 months (16)
* NIRS assessment including: number of blocks/region of interest, block hemogram value, block hemogram colors [red (p < 0.57), orange (0.57 ≤ p < 0.84), tan (0.84 ≤ p < 0.98) and yellow (p ≥ 0.98)]. (20)
* IVUS assessment including: mean lumen area (mm2), mean vessel area (mm2), mean scaffold area (mm2), mean plaque area (mm2), plaque volume (mm3), calcification volume (mm3), hyperechogenicity (mm3 and %).
* Coronary response expressed as percent change from baseline of the acetylcholine- and nitroglycerine-induced change in mean lumen diameter.
* Device-oriented composite end-point as defined by Academic Research Consortium, consisting of cardiac death, myocardial infarction (not clearly attributable to a non-target vessel), target lesion revascularization at 6, 18 and 36 months. (21)
* Patient-oriented composite end-point as defined by Academic Research Consortium, consisting of all-cause mortality, any myocardial infarction (including non-target vessel territory) and repeat revascularization (includes all target and nontarget vessel) at 6, 18 and 36 months. (21)
* Quality of life assessed by generic and specific cardiology psychology tools (QLI, MacNew, EQ-5D) validated in coronary artery disease patients (especially related to angina) at 6, 18 and 36 months.

Study design

The study will assess the safety and performance of the Fantom sirolimus eluting BVS in the acute setting of myocardial infarction with unstable lesions and thrombogenic milieu.

This is a prospective evaluation of clinical and patient related measures in STEMI patient who undergo urgent primary percutaneous coronary intervention (PCI) with stent implantation. Patients with culprit lesions with 2.5 - 3.5 mm diameter and located in one of the main coronary arteries will be included in the trial and prospectively observed. The study will comprise 20 patients, who will undergo additional evaluation with OCT and NIRS/IVUS at baseline, 6 months, 18-24 months and 36 months.

The device will be delivered in sizes 2.5 and 3.0 in diameter / 18 and 24 mm and 3.5 mm x 18 mm in length.

Patient population

Total of 20 STEMI patients will be enrolled in this study.

Patient eligibility

The FANTOM STEMI trial will include individuals with confirmed electrocardiographic and angiographic diagnosis of STEMI, who are eligible for BVS implantation during the primary PCI. Only patients who sign informed consent and meet all of the inclusion and none of the exclusion criteria will be enrolled in the study. The final decision regarding inclusion will be taken after lesion preparation and intravascular imaging assessment.

Inclusion criteria

Candidates must meet ALL of the following inclusion criteria:

* Electrocardiographic confirmation of acute coronary syndrome with ST segment elevation (according to the 2012 European Society of Cardiology guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation) or high-risk non-ST segment elevation patients in whom urgent reperfusion strategy is applied.
* Symptom onset to balloon inflation time <12 hours
* Age >18 years
* The patient's written informed consent has been obtained prior to the procedure.
* Each lesion must meet all the following baseline criteria (prior to pre-dilation):

  * De novo lesion in a native coronary artery.
  * Visually estimated stenosis of at least 50%.
  * Visually estimated RVD ≥2.5 mm and ≤3.5 mm (RVD defined as mean of proximal and distal RVD)
  * Lesion length:

    * 20 mm by visual estimate for single scaffold implantation
* Each lesion must meet all the following criteria after pre-dilatation:

  * Target vessel reference diameter ≤3.5 mm by visual assessment.
  * Lesion length:

    * 20 mm by visual estimate for single scaffold implantation

Exclusion criteria

Candidates will be excluded from the trial if ANY of the following exclusion criteria are met:

A. Clinical

* Cardiogenic shock or pulmonary edema
* Known hypersensitivity or contraindication to acetylsalicylic acid, clopidogrel, prasugrel, ticagrelor, heparins, abciximab, everolimus, or polylactide
* Hypersensitivity to contrast agents
* Concomitant diseases resulting in significantly worse long-term prognosis
* Acute and chronic inflammatory conditions
* Lack of patient consent
* Acute mechanical complications of myocardial infarction
* Known pregnancy at time of randomization. Female who is breastfeeding at time of randomization.
* Fibrinolysis prior to PCI.
* Active bleeding or coagulopathy or patient at chronic anticoagulation therapy
* Life expectancy less then 12 months.
* Patient has a scheduled surgery or another contraindications that may preclude 12-month dual antiplatelet therapy.
* Subject participating in an other trial B. Angiographic
* Significant left main coronary artery stenosis
* Multivessel disease requiring coronary artery bypass grafting (MVD scheduled for percutaneous treatment is not considered as an exclusion criteria).
* Culprit lesion location within a true bifurcation with a large side branch (vessel lumen diameter >2.0 mm)
* Presence of massive calcifications seen within the vessel contour or identified using intracoronary imaging techniques
* Lesion within a vein bypass graft
* Lesions located within 3 mm from vessel origin
* Target lesion located within previously stented region
* Anatomic location and lesion morphology precluding an optimal effect of percutaneous coronary intervention (PCI) or imaging by OCT in the opinion of the investigator
* Excessive proximal tortuosity
* Vessel diameter <2.5 mm and > 3.5 mm

Study procedure

Screening procedure

All patient who are admitted to the study site will be evaluated based on this protocol with intention for study inclusion (patient screening). All patients with STEMI will be considered as potentially eligible candidates. Before being approach with patient informed consent (PIC), the member of study team will explain all the risks and benefits associated with the procedure and allow enough time to the patient for asking any questions that might represent his/her concerns. The patient must sign the consent prior to enrollment; failure to do so is a subject for ineligibility. After PIC is acquired, the patient will receive a unique screening number consisting of three digits (i.e. 001).

The initial evaluation comprises of the following elements:

* History of symptoms directly leading to the diagnosis
* Cardiac physical examination
* 12-lead ECG
* Coronary angiogram.

Thereafter, all inclusion and exclusion criteria will be rechecked. If not all inclusion criteria are met, or there are at least one-exclusion criteria present the patient will be considered as screening failure.

Patient allocation

All patient who meet all eligibility criteria after pre-dilatation will be allocated in the study and have a Fantom BVS implanted.

Medications

Pre-treatment

The pretreatment with aspirin, P2Y12 inhibitor and heparin is allowed as per local practice. In case the patient did not receive all of the above-mentioned drugs, those will be administered in latest just after coronary angiogram. The desired doses are: aspirin of 300 mg p.o., P2Y12 inhibitor according to the agent (600 mg of clopidogrel or 60 mg of prasugrel or 180 mg of ticagrelor), and unfractionated heparin of 70-100 units per kg (or 50-60 units per kg, if IIb/IIIa inhibitor if co-administered).

Peri-procedural

If no anticoagulant was administered in the pre-hospital setting an intravenous agent should be given in the cathlab (preferably UFH). If UFH is used, the anticoagulation should be monitored according to the activated clotting time > 250 second (200-250 seconds if GP IIb/IIIa inhibitor is being administered). The GP IIb/IIIa inhibitors may be administered at operator discretion. Before final angiographic projections, the nitroglycerin should be administered i.c.

Post-procedural

After the procedure patients should be treated according to the European Society of Cardiology Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation. Dual antiplatelet therapy (DAPT) must me maintained for consecutive 12-months after revascularization comprising of low dose aspirin (75-100 mg daily) and a maintenance dose of P2Y12 inhibitor (clopidogrel 75 mg daily, prasugrel 10 mg daily, ticagrelor 90 mg bid). In patients with an indication to long-term anticoagulation the length of DAPT should be adjusted according to individual risk factors.

All patients should receive optimal medical therapy consisting of high dose statins, additionally in those with low ejection fraction beta-blockers, angiotensin converting enzyme inhibitors, and aldosterone antagonists should be considered if not contraindicated.

ELIGIBILITY:
Inclusion Criteria:

* • Electrocardiographic confirmation of acute coronary syndrome with ST segment elevation (according to the 2012 European Society of Cardiology guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation) or high-risk non-ST segment elevation patients in whom urgent reperfusion strategy is applied.

  * Symptom onset to balloon inflation time <12 hours
  * Age >18 years
  * The patient's written informed consent has been obtained prior to the procedure.
  * Each lesion must meet all the following baseline criteria (prior to pre-dilation):

    * De novo lesion in a native coronary artery.
    * Visually estimated stenosis of at least 50%.
    * Visually estimated RVD ≥2.5 mm and ≤3.5 mm (RVD defined as mean of proximal and distal RVD)
    * Lesion length:

      * 20 mm by visual estimate for single scaffold implantation
  * Each lesion must meet all the following criteria after pre-dilatation:

    * Target vessel reference diameter ≤3.5 mm by visual assessment.
    * Lesion length:

      * 20 mm by visual estimate for single scaffold implantation

Exclusion Criteria:

Candidates will be excluded from the trial if ANY of the following exclusion criteria are met:

A. Clinical

* Cardiogenic shock or pulmonary edema
* Known hypersensitivity or contraindication to acetylsalicylic acid, clopidogrel, prasugrel, ticagrelor, heparins, abciximab, everolimus, or polylactide
* Hypersensitivity to contrast agents
* Concomitant diseases resulting in significantly worse long-term prognosis
* Acute and chronic inflammatory conditions
* Lack of patient consent
* Acute mechanical complications of myocardial infarction
* Known pregnancy at time of randomization. Female who is breastfeeding at time of randomization.
* Fibrinolysis prior to PCI.
* Active bleeding or coagulopathy or patient at chronic anticoagulation therapy
* Life expectancy less then 12 months.
* Patient has a scheduled surgery or another contraindications that may preclude 12-month dual antiplatelet therapy.
* Subject participating in an other trial B. Angiographic
* Significant left main coronary artery stenosis
* Multivessel disease requiring coronary artery bypass grafting (MVD scheduled for percutaneous treatment is not considered as an exclusion criteria).
* Culprit lesion location within a true bifurcation with a large side branch (vessel lumen diameter >2.0 mm)
* Presence of massive calcifications seen within the vessel contour or identified using intracoronary imaging techniques
* Lesion within a vein bypass graft
* Lesions located within 3 mm from vessel origin
* Target lesion located within previously stented region
* Anatomic location and lesion morphology precluding an optimal effect of percutaneous coronary intervention (PCI) or imaging by OCT in the opinion of the investigator
* Excessive proximal tortuosity
* Vessel diameter <2.5 mm and > 3.5 mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-06-06 (Actual); Primary Completion 2019-06-06 (Estimated); Study Completion 2022-06-06 (Estimated)

PRIMARY OUTCOMES:
Procedural success defined as acute angiographic success (residual stenosis <20% and TIMI flow 3) without in-hospital major adverse cardiac events (MACE) | From time of procedure until the date of discharge from hospital assessed up to 30 days

SECONDARY OUTCOMES:
Angiographic success defined as device implantation into target lesion with residual stenosis of < 20% and presence of grade 3 TIMI flow assessed by angiography | 3 years
Quantitative coronary angiographic measurements including minimum lumen diameter (mm), late lumen loss (mm) evaluated post-procedure at 6, 18 and 36 months | 3 years
OCT measurements at patient level evaluated post-procedure, at 6, 18 and 36 months. | 3 years
Quantitative coronary angiographic measurements including diameter stenosis (%) at 6, 18 and 36 months | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- 1st Department of Cardiology, Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided